CLINICAL TRIAL: NCT04083170
Title: Infusion of Off-the-Shelf Ex Vivo Expanded Cryopreserved Progenitor Cells to Facilitate the Engraftment of a Single CCR5Δ32 Homozygous or Heterozygous Cord Blood Unit in Patients With HIV and Hematological Malignancies
Brief Title: Cord Blood Transplant With Dilanubicel for the Treatment of HIV Positive Hematologic Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The federal funding period ended. The study was originally intended to be multi-site but was only conducted at the lead site. Due to the rarity of the subject population & smaller # of enrolling sites, we were not able to reach accrual goals.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Filippo Milano, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1004070; NCI-2019-05729 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R34HL142322 (NIH); 10304 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Acute Erythroid Leukemia; Acute Lymphoblastic Leukemia; Acute Megakaryoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid Cell Neoplasm; HIV Infection; Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts; Non-Hodgkin Lymphoma; Refractory Anemia
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Neoplasms; HIV Infections; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Anemia, Refractory | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Thiotepa; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (fludarabine, cyclophosphamide, TBI, dilanubcel) (Experimental): Patients receive fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6, and undergo TBI BID on days -4 to -1. Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation; Biological: Dilanubicel
- Regimen B (anticancer drugs, TBI, dilanubicel) (Experimental): Patients receive fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo TBI QD on days -2 to -1. Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Thiotepa; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation; Biological: Dilanubicel

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: 118218; 2-Fluoro-9-beta-arabinofuranosyladenine; 2-Fluorovidarabine; 9-Beta-D-arabinofuranosyl-2-fluoroadenine; Fluradosa
Drug: Cyclophosphamide — Given IV
  Other Names: Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan
Drug: Thiotepa — Given IV
  Other Names: STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thiofosfamide; Thio-Tepa; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; Triethylene thiophosphoramide; Triethylenethiophosphoramide; TSPA; WR 45312
  Arms: Regimen B (anticancer drugs, TBI, dilanubicel)
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; TOTAL BODY IRRADIATION; Whole Body Irradiation; Whole-Body Irradiation; SCT_TBI
Procedure: Umbilical Cord Blood Transplantation — Undergo UCBT
  Other Names: Cord Blood Transplantation; UCB transplantation
Biological: Dilanubicel — Given IV
  Other Names: Allogeneic UCB-derived Hematopoietic Stem and Progenitor Cells NLA101; Allogeneic Umbilical Cord Blood-derived HSPCs NLA101; NLA101

SUMMARY:
This phase II trial studies the side effects of a cord blood transplant using dilanubicel and to see how well it works in treating patients with human immunodeficiency virus (HIV) positive hematologic (blood) cancers. After a cord blood transplant, the immune cells, including white blood cells, can take a while to recover, putting the patient at increased risk of infection. Dilanubicel consists of blood stem cells that help to produce mature blood cells, including immune cells. Drugs used in chemotherapy, such as fludarabine, cyclophosphamide, and thiotepa, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Total body irradiation is a type of whole-body radiation. Giving chemotherapy and total-body irradiation before a cord blood transplant with dilanubicel may help to kill any cancer cells that are in the body and make room in the patient's bone marrow for new stem cells to grow and reduce the risk of infection.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 2 regimens.

REGIMEN A: Patients receive fludarabine intravenously (IV) over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6, and undergo total body irradiation (TBI) twice daily (BID) on days -4 to -1. Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.

REGIMEN B: Patients receive fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo TBI once daily (QD) on days -2 to -1. Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28, 80, and 180 days, and then at 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* >= 6 months to =< 65 years
* Treatment with combination antiretroviral therapy (cART) for at least 1 month before enrollment
* Viral load < 5000 copies/ml plasma on cART
* Disease criteria

  * Acute myeloid leukemia

    * High risk in first complete remission (CR1), >= 2 cycles to obtain complete remission (CR), erythroblastic or megakaryocytic leukemia; >= in second complete remission (CR2)
    * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%
    * Patients for whom adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible. Specimen for morphologic assessment, including possible repeat procedures will be obtained (as possible). These patients must be discussed with the lead principal investigator, Filippo Milano prior to enrollment
  * Acute lymphoblastic leukemia

    * High risk CR1 (for example, but not limited to: t(9;22), t(1;19), t(4;11) or other mixed-lineage leukemia [MLL] rearrangements, hypodiploid); greater than 1 cycle to obtain CR; >= CR2
    * All patients must be in CR as defined by hematologic recovery and < 5% blasts by morphology within the bone marrow and a cellularity of >= 15%
    * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible. Specimen for morphologic assessment, including possible repeat procedures will be obtained (as possible). These patients must be discussed with the lead principal investigator, Filippo Milano prior to enrollment
  * Chronic myelogenous leukemia excluding refractory blast crisis. To be eligible in first chronic phase (CP1) patient must have failed or be intolerant to imatinib mesylate
  * Myelodysplasia (MDS) International Prognostic Scoring System (IPSS) intermediate (Int)-2 or high risk (i.e., refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation [RAEBt]) or refractory anemia with severe pancytopenia or high-risk cytogenetics. Blasts must be < 10% by a representative bone marrow aspirate morphology
  * Other hematologic malignancy such as non-Hodgkin lymphomas. Fred Hutch site: These patients must be presented at Patient Care Conference (PCC) prior to enrollment, given potential competing eligibility on auto-transplant protocols. Participating centers: These patients must be discussed with the lead principal investigator, Filippo Milano prior to enrollment
* Karnofsky (>= 16 years old) >= 70%
* Lansky (< 16 years old) >= 50%
* Adults: Calculated creatinine clearance must be > 60 mL and serum creatinine =< 2 mg/dL
* Children (< 18 years old): Calculated creatinine clearance must be > 60 mL/min
* Total serum bilirubin must be < 3 mg/dL
* Transaminases must be < 3 x the upper limit of normal
* Diffusion capacity of the lung for carbon monoxide (DLCO) corrected > 50% normal or for pediatric patients in whom DLCO cannot be measured has adequate pulmonary function
* Left ventricular ejection fraction > 45% OR
* Shortening fraction > 26%
* Ability to understand and the willingness to sign a written informed consent document (adult subject or parent/legal guardian of minor subject)

Exclusion Criteria:

* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* Pregnant or breastfeeding
* Prior myeloablative transplant within the last 6 months
* Extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation
* Central nervous system (CNS) leukemic involvement not clearing with intrathecal chemotherapy. Diagnostic lumbar puncture to be performed

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Milano, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Cord Blood Center, Cleveland, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel): Patients receive fludarabine IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6, and undergo TBI BID on days -4 to -1 (totaling 1320 cGy). Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.
  Fludarabine: Given IV
  Cyclophosphamide: Given IV
  Total-Body Irradiation: Undergo TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT
  Dilanubicel: Given IV
- Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel): Patients receive fludarabine IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo TBI QD on days -2 to -1 (totaling 400 cGy). Patients then undergo umbilical cord blood transplant on day 0. Between 4-24 hours after transplant completion, patients receive dilanubicel IV over 5-10 minutes in the absence of disease progression or unacceptable toxicity.
  Fludarabine: Given IV
  Cyclophosphamide: Given IV
  Thiotepa: Given IV
  Total-Body Irradiation: Undergo TBI
  Umbilical Cord Blood Transplantation: Undergo UCBT
  Dilanubicel: Given IV
Period: Overall Study
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants enrolled to Regimen A of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] |  | 21 [21 to 21] | 21 [21 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 1 | 1
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
Matched cord blood unit with either homozygous or heterozygous CCR5Δ32 mutation. [Count of Participants; unit: Participants]
  Homozygous CCR5Δ32 Mutation in CBU |  | 1 | 1
  Heterozygous CCR5Δ32 Mutation in CBU |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Graft Failure Rejection
Description: Will be defined by no neutrophil recovery by day 45 (regardless of donor chimerism) or autologous recovery (neutrophil recovery but < 10% donor chimerism in blood and bone marrow) by day 36. This outcome was originally intended to be assessed for per the aforementioned definitions, but was only able to be assessed through 35 days post-transplant.
Time Frame: Up to day 35 post-transplant
Population: No participants were enrolled to Regimen A of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Dilanubcel) | Regimen B (Anticancer Drugs, TBI, Dilanubicel)
Number analyzed (Participants) | 0 | 1
Participants |  | 0

2. Secondary Outcome: Incidence of Infusion Toxicities
Description: Defined as Common Terminology Criteria for Adverse Events version 5.0 grade >= 3 events.
Time Frame: Within the first 24 hours after infusion
Population: No participants were enrolled to Regimen A of the study.
Measure: Number; unit: infusion toxicity events
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
infusion toxicity events |  | 0

3. Secondary Outcome: Median Number of Days Post-Transplant to Neutrophil Recovery Occurred
Description: Neutrophil recovery is defined as the first day of 2 consecutive days of absolute neutrophil count >= 500 after the first post-cord blood transplant nadir. This outcome was originally intended to be assessed for up to 45 days post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: Up to Day 35 post-transplant
Population: No participants were enrolled to Regimen A of the study.
Measure: Median (Full Range); unit: Days post-transplant
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
Days post-transplant |  | 16 [16 to 16]

4. Secondary Outcome: Platelet Engraftment
Description: Will be defined as the first day of a platelet count > 20,000/ul with subsequent transfusions for 7 days. This outcome was originally intended to be assessed for up to 2 years post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: 35 days post-transplant
Population: No participants were enrolled to Regimen A of the study. The single Regimen B participant did not achieve platelet engraftment prior to death on Day +35 post-transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
Participants |  | 0

5. Secondary Outcome: Incidence of Severe (Grades III-IV) Acute Graft Versus Host Disease (GVHD)
Description: Will be defined by the 2014 National Institutes of Health (NIH) criteria. This outcome was originally intended to be assessed for up to 2 years post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: 35 days post-transplant
Population: No participant was enrolled to Regimen A of the study.
Measure: Number; unit: Number of Grade 3/4 aGVHD Events
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
Number of Grade 3/4 aGVHD Events |  | 0

6. Secondary Outcome: Incidence of Chronic GVHD
Description: Will be defined by the 2014 NIH criteria. This outcome was originally intended to be assessed for up to 2 years post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: 35 days post-transplant
Population: No participants were enrolled to Regimen A of the study.
Measure: Number; unit: Number of cGVHD Events
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
Number of cGVHD Events |  | 0

7. Secondary Outcome: Incidence of Non-relapse Mortality
Description: Will be defined as death without a prior relapse. This outcome was originally intended to be assessed for up to 180 days post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: 35 days post-transplant
Population: No participants were enrolled to Regimen A of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
Participants |  | 1

8. Secondary Outcome: Human Immunodeficiency Virus (HIV) Plasma Viral Load
Description: Assess CCR5Δ32 cord blood stem cell engraftment and its effect on biomarkers of HIV-1 infection, including plasma viral load and replication-competent reservoirs, as well as in gut and other sites (if tissue samples are available). This outcome was originally intended to be assessed weekly for up to 2 years post-transplant, but was only able to be assessed through 35 days post-transplant.
Time Frame: Baseline and weekly to 35 days post-transplant
Population: No participants were enrolled to Regimen A of the study.
Measure: Number; unit: percentage of viral load change
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 1
percentage of viral load change |  | 0

9. Secondary Outcome: Immune Homeostasis
Description: Concentration of immunity cells per microliters after transplant
Time Frame: Up to 2 years
Population: No participants survived until 2 years, so outcome could not be measured.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Immune Reconstitution
Description: Concentration of immunity cells per microliters after transplant
Time Frame: Up to 2 years
Population: No participants survived until 2 years, so outcome could not be measured.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in HIV-1 Induced Inflammatory Immune Responses
Description: HIV viral load by PCR (copies per milliliter; mL)
Time Frame: Up to 2 years
Population: No participants survived until 2 years, so outcome could not be measured.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: HIV Rebound Following Antiretroviral Therapy (ART) Cessation
Description: Count of participants with HIV rebound, measured by HIV viral load by PCR (copies per milliliter; mL)
Time Frame: Up to 2 years
Population: No participants survived until 2 years, so outcome could not be measured.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Viral Kinetics Following ART Cessation
Description: HIV viral load by PCR (copies per milliliter; mL)
Time Frame: Up to 2 years
Population: No participants survived until 2 years, so outcome could not be measured.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed from start of conditioning until participant death on study at Day 35 post-transplant.
Description: Adverse events were routinely assessed via standard of care clinic visits with laboratory assessments.
Arm/Group | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel)
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) (N=0) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) (N=1)
Hepatobiliary disorders - Other, Liver insufficiency (Hepatobiliary disorders) | 0 | 1 (1) — Liver insufficiency
Renal and urinary disorders - Other, Renal insufficiency (Renal and urinary disorders) | 0 | 1 (1) — Renal insufficiency
Posterior Reversible Encephalopathy Syndrome (PRES) (Nervous system disorders) | 0 | 1 (1) — PRES
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Fludarabine, Cyclophosphamide, TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) (N=0) | Regimen B (Anti-cancer Drugs Plus TBI, Followed by Unmanipulated Cord Blood and Dilanubicel) (N=1)
Sepsis (Strep mitis + Strep salivarius + Staph sp.) (Infections and infestations) | 0 | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 | 1 (1)
Acute kidney injury (AKI) (Renal and urinary disorders) | 0 | 1 (1) — AKI
Myocardial infarction (Cardiac disorders) | 0 | 1 (1)

LIMITATIONS AND CAVEATS:
The study was originally intended to be multi-site but ended up only being conducted at the lead site. Due to the rarity of the subject population and the smaller number of enrolling sites, we were not able to reach accrual goals. Once the funding period ended, the study had to be closed to accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT04083170/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04083170/ICF_000.pdf